CLINICAL TRIAL: NCT04994457
Title: Patient Performance on Virtual Reality Visual Field Devices as Compared to Standard of Care
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Elena Bitrian, Associate Professor of Clinical, University of Miami
Other Study IDs: 20210472
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma
Keywords: Visual Field; Virtual Reality
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Adults with Glaucoma or Suspected Glaucoma: Adults with Glaucoma or Suspected Glaucoma, who have previously had standard automated perimetry (SAP) and will receive virtual reality visual field (VRVF) as part of the standard of care
  Interventions: Device: Virtual Reality Visual Field
- Visual Field Naive Adults: Visual Field Naive Adults will receive SAP and VRVF
  Interventions: Device: Virtual Reality Visual Field; Diagnostic Test: Standard Automated Perimetry
- Children with Glaucoma or Suspected Glaucoma: Children with Glaucoma or Suspected Glaucoma, who have previously had SAP and will receive VRVF as part of the standard of care
  Interventions: Device: Virtual Reality Visual Field
- Visual Field Naive Children: Visual Field Naive Children will receive SAP and VRVF
  Interventions: Device: Virtual Reality Visual Field; Diagnostic Test: Standard Automated Perimetry
- Remote Care Arm: Glaucoma or Suspected Glaucoma participants, who have previously had SAP and will receive VRVF at their home
  Interventions: Device: Virtual Reality Visual Field
- Ptosis Arm: Patients diagnosed with Ptosis, brow ptosis, or dermatochalasis, will receive a specialized version of VRVF and SAP, specifically to detect ptosis
  Interventions: Device: Virtual Reality Visual Field; Diagnostic Test: Standard Automated Perimetry

INTERVENTIONS:
Device: Virtual Reality Visual Field — A head-mounted perimeter with a wireless remote connected to a laptop that monitors responses
Diagnostic Test: Standard Automated Perimetry — Standard of care perimeter
  Groups: Ptosis Arm; Visual Field Naive Adults; Visual Field Naive Children

SUMMARY:
The purpose of this research is to study the effectiveness and patient experience when measuring visual fields using virtual reality goggles.

ELIGIBILITY:
Inclusion:

* Any individual who is physically able to take a virtual reality visual field test
* Patients who either have glaucoma, are glaucoma suspects, or have a strong family history of glaucoma, or have other visual field defects, and normal individual
* Age: Individuals who are old enough to comprehend the instructions and procedures (1-90)

Exclusion:

* Adults unable to consent, prisoners
* Participants who are too tired to take a visual field test
* Participants who refuse to consent
* Individuals who are functionally unable to use VRVF

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are glaucoma or glaucoma suspect who are being seen at Bascom Palmer Eye Institute and/or healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity of VRVF compared to SAP | Day 1
  Sensitivity of VRVF will be determined by comparing Hodapp Anderson Parrish (HAP) Scores, which assess the severity of visual field defects, to those of SAP
Specificity of VRVF compared to SAP | Day 1
  Specificity of VRVF will be determined by comparing Hodapp Anderson Parrish (HAP) Scores, which assess the severity of visual field defects, to those of SAP

SECONDARY OUTCOMES:
Variability of Mean Deviation | Day 1
  Variability of the mean deviation scores obtained from VRVF and SAP

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bitrian, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLaughlin DE, Savatovsky EJ, O'Brien RC, Vanner EA, Munshi HK, Pham AH, Grajewski AL. Reliability of Visual Field Testing in a Telehealth Setting Using a Head-Mounted Device: A Pilot Study. J Glaucoma. 2024 Jan 1;33(1):15-23. doi: 10.1097/IJG.0000000000002290. Epub 2023 Aug 14. PMID 37647317